CLINICAL TRIAL: NCT00556166
Title: Enterra Therapy Gastric Stimulation System
Acronym: Enterra
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal investigator left institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA5072
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Gastroparesis
Keywords: Enterra therapy; Gastric Simulation System
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enterra Therapy (Experimental): The Enterra Therapy Gastric Stimulator will be used on subjects who have failed all other medical options to treat gastroparesis and all have a gastric stimulator implanted.
  Interventions: Device: Enterra Therapy Gastric Stimulator

INTERVENTIONS:
Device: Enterra Therapy Gastric Stimulator — The intramuscular stomach leads, implanted in a minimally invasive surgical procedure lasting 1-3 hours, are placed on the greater curvature of the stomach. The implanted pulse generator (IPG) is about 2 1/2" x 2" x 1/2" and is implanted in a subcutaneous pocket, generally created in the abdominal area, and is then connected to the leads. The IPG provides the energy source that delivers the electrical pulse to the stomach muscle through the stomach leads to improve the symptoms of gastroparesis.
  The doctor will use an external programmer to change the settings of the neurostimulator and control the neurostimulator after implantation. Part of the programmer is held outside the body over the implant site and can adjust or change the settings of the neurostimulator using radio remote control.

SUMMARY:
Enterra Therapy Gastric Simulation System (Enterra Therapy) is indicated for the treatment of patients with long term, uncontrolled (not helped by medication) nausea and vomiting from gastroparesis of diabetic or idiopathic origin.

In March 2000, the Food and Drug Administration (FDA) gave approval of a humanitarian Device Exemption (HDE) of a Humanitarian Use Device (HUD) for Enterra Therapy Gastric electrical (GES) Simulation System. Although, there is evidence that suggests the use of Enterra Therapy System probably helps patients, symptoms, the FDA's HDE approval indicates that the helpfulness of this therapy has not been proven. Physicians at Columbia University Medical Center hope to prove the helpfulness of this device.

DETAILED DESCRIPTION:
Gastroparesis is a debilitating disease in which patients suffer from a number of upper gastrointestinal (GI) symptoms including nausea, vomiting, early satiety, bloating, postprandial fullness, epigastric pain and burning, and cardiac pain and burning. Severe symptoms, particularly vomiting and nausea, can significantly impair a patients daily activities and quality of life.

Current medical practice for the treatment and/or management of gastroparesis consists of dietary modifications, drug therapies, enteral feeding, parenteral feeding and surgery. These treatments are successful for some patients, but have significant drawbacks. Patients may initially be treated with various dietary modifications including frequent low fat meals. However, if dietary modifications alone are unsuccessful, antiemetic and prokinetic drugs, or combinations thereof, are generally tried. If symptoms cannot be controlled with medication, supplemental nutrition via enteral or parenteral feeding may be required to maintain hydration and nutritional status. Prokinetic drugs are intended to promote gastric motility, i.e., to return abnormally slow gastric emptying states to normal. Antiemetic drugs are intended to alleviate symptoms of nausea and vomiting, but have no effect on motility. None of the prokinetic drugs are labeled for improved gastric emptying in gastroparesis. Metoclopramide is the only antiemetic or prokinetic drug indicated for use in the treatment of symptoms of diabetic gastroparesis.

Surgical procedures are occasionally employed to manage symptoms of gastroparesis while maintaining the ability for enteral feeding. Surgical procedures, including gastrectomy, pyloroplasty, and gastrojejunostomy, have had limited success in managing symptoms of gastroparesis. When drug therapies or surgery are ineffective, supplemental enteral feeding via gastric or jejunal feeding tubes or total parenteral nutrition (TPN) may be required to meet the patient's nutritional needs.

For those patients who cannot be adequately treated or managed by current medical practice, the GES has no satisfactory alternative. It is this group of patients for which the GES System is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic(long term, lasting greater than 3 months)
* Intractable (drug refractory, failed medical management with prokinetic and antiemetic drugs
* Failed dietary modifications, and/or requiring enteral feeding) nausea and vomiting secondary to gastroparesis of diabetic or idiopathic etiology

Exclusion Criteria:

* Only patients whom the physician determines are not a candidate for surgical procedures and/or anesthesia due to physical or mental conditions will be excluded. This includes pregnant women, anyone unable to tolerate general anesthesia, and uncorrectable coagulopathy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L. Fowler, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No data available to share as the PI left the institution before the study could finish.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enterra Therapy
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enterra Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Non-specific gender count | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Episodes of Nausea and Vomiting
Description: Data was not analyzed because PI left institution and terminated the study early.
Time Frame: 1 year
Arm/Group | Enterra Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Episodes of Abdominal Pain, Bloating, and Early Satiety
Description: Data was not analyzed because PI left institution and terminated the study early.
Time Frame: 1 year
Arm/Group | Enterra Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Enterra Therapy
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes